CLINICAL TRIAL: NCT03625063
Title: Investigation of Pulmonary Rehabilitation on Exercise Capacity, Physical Activity Level, Respiratory Muscle Strength and Endurance During Transplantation Process in Hematopoietic Stem Cell Transplantation Recipients
Brief Title: Effects of Pulmonary Rehabilitation in Hematopoietic Stem Cell Transplantation Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Gazi University 8
Record Dates: First submitted 2018-07-19; First posted 2018-08-10 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: exercise capacity; physical activity; respiratory muscle strength; respiratory muscle endurance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training group (Active Comparator): Inspiratory muscle, upper extremity aerobic exercise and progressive resistance trainings
  Interventions: Other: Exercise training group
- Control training group (Sham Comparator): Upper extremity aerobic exercise and progressive resistance trainings
  Interventions: Other: Control training group

INTERVENTIONS:
Other: Exercise training group — All exercise program will be applied during supervised session by a physiotherapist. Range of maximal heart rate will be screened by heart rate monitor during supervised session each day at patient's room. Inspiratory muscle training (threshold loading device (Threshold®- Inspiratory Muscle Trainer) at 20-30% of maximal inspiratory pressure (MIP)), upper extremity aerobic exercise training (arm ergometer, at 60-80% of maximum heart rate, dyspnea perception at 3-4 level as well as fatigue perception at 5-6 level according to Modified Borg Scale) and progressive resistance training (shoulder flexors, shoulder abduction and knee extensors at 4-6 level according to modified Borg scale) will be performed in the treatment group during acute hematopoietic stem cell transplantation process.
  Arms: Exercise training group
Other: Control training group — All exercise program will be applied during supervised session by a physiotherapist. Range of maximal heart rate will be screened by heart rate monitor during supervised session each day in patient's room.Upper extremity aerobic exercise training (arm ergometer, at 60-80% of maximum heart rate, dyspnea perception at 3-4 level as well as fatigue perception at 5-6 level according to Modified Borg Scale) and progressive resistance training (shoulder flexors, shoulder abduction and knee extensors at 4-6 level according to modified Borg scale) except inspiratory muscle training will be performed in the control group during acute hematopoietic stem cell transplantation process.
  Arms: Control training group

SUMMARY:
Stem cell transplantation is a process in which stem cells are harvested from either a patient's or donor's bone morrow or peripheral blood for intravenous infusion. Hematopoietic stem cell transplantation is a treatment with a high curative potential that may benefit a great number of patients with hematological, oncological, immunologic and hereditary diseases. In contrast, there are significant risks of chronic and acute complications due to conditioning regimens and immunosuppression, toxicity infections, graft versus host disease (GVHD) and inactivity including being bedridden. Patients undergoing hematopoietic stem cell transplantation are exposed to risk factors due to chemotherapy, whole body radiation, high dose corticosteroids, treatment-related inactivity, transplantation and GVHD-related muscle damage. Direct toxicity of the cardiovascular and musculoskeletal system (left ventricular dysfunction, pulmonary fibrosis) in relation to hematopoietic stem cell transplantation and secondary indirect physiological consequences of treatment such as exercise intolerance, sarcopenia are seen.

In literature, there are few studies showing that aerobic exercise and resistance training applied during and after the transplantation process has positive effects on muscle strength and endurance, fatigue, functional performance, quality of life and physical activity. It has been shown in the literature that inspiratory muscle training in allogeneic hematopoietic stem cell transplant recipients increases functional exercise capacity, inspiratory and expiratory muscle strength, and reduces effort dyspnea perception, but the effects of inspiratory muscle training during transplantation have not been investigated. There are no studies showing long-term follow-up of comprehensive cardiopulmonary rehabilitation program during hematopoietic stem cell transplantation and which of these outcome measures are survival effect. Therefore, the investigators aimed to investigate the effect of cardiopulmonary rehabilitation on hematopoietic stem cell transplantation in terms of exercise capacity, respiratory and peripheral muscle strength, respiratory muscle endurance, respiratory function, physical activity level, fatigue, depression and quality of life effects and the effect of these outcome measures on survival.

DETAILED DESCRIPTION:
According to sample size calculation 20 patients scheduled for hematopoietic stem cell transplantation will be included. Patients scheduled for hematopoietic stem cell transplantation will be evaluated four times; pre-transplantation, post-transplantation, 100th day after transplantation and 1st year after transplantation. Recipients will be randomized into study and control groups. Cardiopulmonary rehabilitation programme includes inspiratory muscle training, upper extremity aerobic exercise, progressive resistance training will be performed study groups. Upper extremity aerobic exercise and progressive resistance training will be performed control groups. Exercise capacity, physical activity, pulmonary functions, respiratory and peripheral muscle strength, respiratory muscle endurance, dyspnea and fatigue perception, depression and quality of life will be evaluated. Primary outcome measurements are exercise capacity and which outcome measures influence survival. Secondary outcomes are respiratory and peripheral muscle strength, respiratory muscle endurance, pulmonary functions, physical activity, dyspnea and fatigue perception, depression and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo hematopoietic stem cell transplantation
* under standard medications
* 18-65 years of age

Exclusion Criteria:

* orthopedic or neurological disease with a potential to affect functional capacity,
* comorbidities such as asthma, chronic obstructive pulmonary disease (COPD), acute infections or pneumonia,
* have problems that can prevent evaluation,
* take treatment other than standard medications during transplantation,
* having acute hemorrhage in the intracranial and / or lung and other areas
* having any contraindication to exercise training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Maximal exercise capacity | Second day
  Maximal exercise capacity will be evaluated symptom limited cardiopulmonary exercise testing. Oxygen consumption will be measured by cardiopulmonary exercise test. The cardiopulmonary exercise test will be performed on the treadmill at a progressively increasing speed and grade.

SECONDARY OUTCOMES:
Respiratory muscle strength | First day
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device .
Respiratory muscle endurance | First day
  It will be evaluated incremental threshold loading test, in which participants started an initial load of 30% of maximal inspiratory pressure with a 10% increment every 2 minutes.
Peripheral muscle strength | First day
  Shoulder abduction and knee extensor muscle strength using portable hand held dynamometer, hand grip strength using grip dynamometer will be evaluated.
Pulmonary functions contains dynamic lung volumes | First day
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria.
  Forced expiratory volume in the first second (FEV1, (liter)) and (FEV1 (%)) , forced vital capacity (FVC (L)) and (FVC (%)), forced expiratory volume in the first second/forced vital capacity (FEV1/FVC (%)) , peak expiratory flow (PEF(L)), and (PEF (%)), and forced expiratory flow from 25 to 75 % (FEF25-75 %(L)), and (FEF25-75 % (%)) will be expressed as the liter and percentages of the predicted values.
Physical activity | First day
  Physical activity will be evaluated multi sensor activity monitor for 4 consecutive days.
Fatigue | First day
  Fatigue Severity Scale (Turkish version) - Fatigue Severity Scale (FSS) is a self-reported questionnaire. FSS evaluates patient's fatigue severity. This questionnaire includes 9 items and score range for each item from 1 to 7 point (7-point Likert scale). Fatigue Severity Scale score is calculates by deriving an arithmetic mean. Cut-scores of over 4 are indicative of significant fatigue (higher scores show more severe fatigue).
Depression | Second day
  Beck Depression Inventory (Turkish version) - Beck Depression Inventory (BDI) is a self-reported questionnaire. BDI evaluates patients' depression level. This questionnaire includes 21 items. Each item scores from 0 to 3 point (higher scores shows patient ). The BAI scores are classified as "depression" over 17 points.
Survival | 100th day and first year
  Kaplan-meier survival analysis will be calculated at 100th day and first year.
Functional exercise capacity | First day
  Functional exercise capacity will be evaluated with 6-minute walking test according to the ATS and ERS criteria.
Disease Specific Quality of Life | First day
  Quality of life was measured using Turkish version of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version 3.0 (EORTCQLQ) which is widely used as health related quality of life questionnaire in cancer patients. The cancer-specific questionnaire has 30 questions and incorporates five functional scales, three symptom scales, a global health status and several single items. All item scores are transformed to 0-100. Higher values indicate higher functional/healthy level in functional scales, a higher quality of life level in global health status and increased symptoms in symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Selin Bayram, MSc, Study Chair — Gazi University; Meral Boşnak Güçlü, Assoc. Prof, Study Director — Gazi University; Gülşah Barğı, PhD, Principal Investigator — Gazi University; Zeliha Çelik, MSc, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelsey CR, Scott JM, Lane A, Schwitzer E, West MJ, Thomas S, Herndon JE 2nd, Michalski MG, Horwitz ME, Hennig T, Jones LW. Cardiopulmonary exercise testing prior to myeloablative allo-SCT: a feasibility study. Bone Marrow Transplant. 2014 Oct;49(10):1330-6. doi: 10.1038/bmt.2014.159. Epub 2014 Jul 28. PMID 25068429
- [Background] Morishita S, Kaida K, Yamauchi S, Wakasugi T, Ikegame K, Ogawa H, Domen K. Relationship of physical activity with physical function and health-related quality of life in patients having undergone allogeneic haematopoietic stem-cell transplantation. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12669. Epub 2017 Feb 21. PMID 28220548
- [Background] Kovalszki A, Schumaker GL, Klein A, Terrin N, White AC. Reduced respiratory and skeletal muscle strength in survivors of sibling or unrelated donor hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 Jun;41(11):965-9. doi: 10.1038/bmt.2008.15. Epub 2008 Feb 11. PMID 18264142
- [Background] Mello M, Tanaka C, Dulley FL. Effects of an exercise program on muscle performance in patients undergoing allogeneic bone marrow transplantation. Bone Marrow Transplant. 2003 Oct;32(7):723-8. doi: 10.1038/sj.bmt.1704227. PMID 13130321
- [Background] Hacker ED, Larson J, Kujath A, Peace D, Rondelli D, Gaston L. Strength training following hematopoietic stem cell transplantation. Cancer Nurs. 2011 May-Jun;34(3):238-49. doi: 10.1097/NCC.0b013e3181fb3686. PMID 21116175
- [Background] Baumann FT, Zopf EM, Nykamp E, Kraut L, Schule K, Elter T, Fauser AA, Bloch W. Physical activity for patients undergoing an allogeneic hematopoietic stem cell transplantation: benefits of a moderate exercise intervention. Eur J Haematol. 2011 Aug;87(2):148-56. doi: 10.1111/j.1600-0609.2011.01640.x. PMID 21545527
- [Background] Bargi G, Guclu MB, Aribas Z, Aki SZ, Sucak GT. Inspiratory muscle training in allogeneic hematopoietic stem cell transplantation recipients: a randomized controlled trial. Support Care Cancer. 2016 Feb;24(2):647-659. doi: 10.1007/s00520-015-2825-3. Epub 2015 Jul 2. PMID 26135532
- [Derived] Bayram S, Bargi G, Celik Z, Bosnak Guclu M. Effects of pulmonary rehabilitation in hematopoietic stem cell transplantation recipients: a randomized controlled study. Support Care Cancer. 2023 Dec 30;32(1):72. doi: 10.1007/s00520-023-08236-x. PMID 38158450